CLINICAL TRIAL: NCT04456621
Title: Proton Beam Radiotherapy for Unresectable Liver Metastasis: Prospective Phase II Trial
Brief Title: Proton Beam Therapy for Unresectable Liver Metastasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Park Hee Chul, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-10-048
Record Dates: First submitted 2020-06-30; First posted 2020-07-02 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Local Control Rate; Side Effect

STUDY DESIGN:
Intervention Model Description: Proton beam radiotherapy : 5 fractions of 12 GyRBE or 10 fractions of 7 GyRBE
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PBT arm (Experimental)
  Interventions: Radiation: PBT

INTERVENTIONS:
Radiation: PBT — Proton beam radiotherapy 70 gray relative biological equivalent (GyRBE)/10 fractions (Fx) or 60 GyRBE/5 Fx

SUMMARY:
The investigators performed the present study to evaluate the role of proton beam therapy for liver metastasis which is unresectable and unsuitable for radiofrequency ablation (RFA) in terms of local control and safety.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed cancer patient
* confirmed liver metastasis via computed tomography (CT) or magnetic resonance imaging (MRI) or biopsy
* unresectable or unsuitable for RFA
* solitary liver metastasis or less than 3 metastatic lesions if the distance is less than 3 cm between metastatic lesions
* case discussed by surgeon, radiologist, and radiation oncologist
* Eastern cooperative oncology group performance status 0 to 2
* optimal liver and renal function (Child-Pugh score 10 or less)
* informed consent
* agree to be contraceptive for the duration of the study and for the next 6 months

Exclusion Criteria:

* uncontrolled ascites or hepatorenal syndrome
* status of pregnancy or breast-feeding
* less than 12 weeks of expected survival
* combined disease known to have high radiation side effects
* serious acute illness that is not treated other than liver disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
6 month local control rate | at the point of 6 month follow-up after proton beam therapy
  local control rate (except local progression)

SECONDARY OUTCOMES:
Overall survival rate | at the point of 2 year follow-up after proton beam therapy
  overall survival rate
6 month side effect | at the point of 6 month follow-up after proton beam therapy
  side effect

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No